CLINICAL TRIAL: NCT03819192
Title: Prediction of Early-Onset Neonatal Sepsis (EONS) in Pregnant Women With Preterm Premature Rupture of Membranes (PPROM) by Vaginal Microbiome Analysis - a Pilot Study
Brief Title: Predicting EONS in PPROM Patients
Acronym: PEONS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jena University Hospital (Other)
Collaborators: Center of Fetal Surgery, University Hospital Halle Saale (Unknown); Section for Neonatology and Pediatric Intensive Care, University Hospital Halle Saale (Unknown)
Responsible Party: Sponsor
Other Study IDs: KG-PEONS
Record Dates: First submitted 2019-01-23; First posted 2019-01-28 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: PPROM; Early-Onset Neonatal Sepsis
MeSH Terms: conditions — Preterm Premature Rupture of the Membranes; Neonatal Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- neonates with signs of EONS
  Interventions: Diagnostic Test: microbiome analysis; Diagnostic Test: Conventional cultures; Diagnostic Test: CAAP48 measurement
- neonates without signs of EONS
  Interventions: Diagnostic Test: microbiome analysis; Diagnostic Test: Conventional cultures; Diagnostic Test: CAAP48 measurement
- pregnant women with PPROM
  Interventions: Diagnostic Test: microbiome analysis; Diagnostic Test: Conventional cultures; Diagnostic Test: CAAP48 measurement

INTERVENTIONS:
Diagnostic Test: microbiome analysis — From all full age pregnant women with PPROM enrolled in this study vaginal smear samples will be taken at three time points:
  1. directly after hospitalization
  2. 5-7 days after beginning of antibiotic treatment
  3. 24 h before birth
  The microbiome of the neonates of these women will be analysed out of pharyngeal and rectal swabs and umbilical cord blood taken directly after birth and additionally out of the first Meconium.
Diagnostic Test: Conventional cultures — For every sample taken for microbiome analysis, a conventional culture is taken as control.
Diagnostic Test: CAAP48 measurement — CAAP48 is an identified sepsis marker in adult patients. The samples are taken dependent on clinical monitoring to compare CAAP48 with established inflammation markers (CRP, IL-6, White blood cell count, Procalcitonin).

SUMMARY:
An EONS occurred in nearly 14-22 % of the preterm infant of pregnant women with PPROM. To this day no risk prediction is established. The main aim of this pilot study is generating primary data with a focus on the vaginal microbiome to set-up a prospective, multi-centre trial investigating the role of the vaginal microbiome for future EONS risk prediction.

The planned PEONS pilot trial is subdivided in three Work packages:

1. Recruitment, sample collection and routine clinical diagnostics
2. Microbiome analysis by 16S rRNA
3. Microbiome/ Metagenome analysis by "Nanopore" (proof-of-principle) and will enroll women with a PPROM event hospitalized between 22+0 and 34+0 weeks of gestation and neonates with signs of EONS (Subgroup 1) and without signs of EONS (Subgroup 2).

ELIGIBILITY:
Inclusion Criteria:

* full age pregnant woman with PPROM and their born preterm infants
* hospitalization between 22+0 and 34+0 weeks of gestation
* multipara possible

Exclusion Criteria:

* hospitalization with PPROM before limit of viability are reached
* intrauterine fetal death
* no study agreement
* not able to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PPROM cohort = PPROM patients (hospitalization between 22+0 - 34+0 weeks of gestation) and their born preterm neonates, n = 65
  * Subgroup 1: with EONS, n = 15
  * Subgroup 2: without EONS, n = 50
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Development of EONS | 3 days after delivery
  Primary outcome is the development of EONS defined as the presence of confirmed or suspected sepsis at ≤3 days after birth for which prolonged neonatal antibiotic treatment beyond 72 hours. Confirmed sepsis is established by positive blood cultures whilst suspected sepsis is diagnosed in the presence of clinical suspicion of sepsis (lethargy, apnoea, respiratory distress, hypotension (mean arterial blood pressure (MAD) < gestational age), hypoperfusion and shock) supported by elevated neonatal C-reactive protein (CRP), interleukin-6 (IL6) or blood film suggestive of bacteraemia.

SECONDARY OUTCOMES:
vaginal CST in PPROM | until delivery
  the specific patterns of vaginal CST and vaginal microbiota composition (microbiome) in PPROM
neonatal microbial colonisation | up to 2 days after delivery
  neonatal microbial colonisation (microbiome) on 1st and 2nd day of life

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - University Hospital Halle/s., Halle, Saxony-Anhalt
  - Jena University Hospital, Jena, Thuringia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dos Anjos Borges LG, Pastuschek J, Heimann Y, Dawczynski K; PEONS study group; Schleussner E, Pieper DH, Zollkau J. Vaginal and neonatal microbiota in pregnant women with preterm premature rupture of membranes and consecutive early onset neonatal sepsis. BMC Med. 2023 Mar 13;21(1):92. doi: 10.1186/s12916-023-02805-x. PMID 36907851